CLINICAL TRIAL: NCT03548766
Title: Using DNA-Typing and Erythrocyte Microparticle Analysis to Detect Homologous/Autologous Blood Doping- a Transfusion Study
Brief Title: Using DNA-Typing and Erythrocyte Microparticle Analysis to Detect Blood Doping
Acronym: Transfusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: World Anti-Doping Agency (Other); Anti-Doping Lab Qatar (Unknown); Sidra Medicine (Other); Laboratorio Antidoping FMSI (Unknown)
Responsible Party: Principal Investigator, Dr. Mohamed A Yassin ,MD, Hematology Consultant, Hamad Medical Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MRC-02-18-070
Record Dates: First submitted 2018-05-06; First posted 2018-06-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Blood Disease; Blood Transfusion, Autologous; Blood Doping; Blood Transfusion, Homologous
MeSH Terms: conditions — Hematologic Diseases | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Subjects (Experimental): Six healthy subjects will receive an ABT (Autologous Blood Transfusion)
  Interventions: Biological: Autologous Blood Transfusion
- Anemic Patients (Experimental): Six patients with anemia will receive a HBT (Homologous Blood Transfusion)
  Interventions: Biological: Homologous Blood Transfusion

INTERVENTIONS:
Biological: Homologous Blood Transfusion — Homologous, or allogenic, blood transfusions involves someone collecting and infusing the blood of a compatible donor into him/herself.
  Other Names: Allogenic Blood Transfusion
  Arms: Anemic Patients
Biological: Autologous Blood Transfusion — Autologous blood transfusion is the collection and re-infusion of the patient's own blood or blood components.
  Arms: Healthy Subjects

SUMMARY:
A total of 12 subjects will be recruited for participation in this study. 6 subjects will receive re-infusion of autologous blood, and 6 subjects (anemic patients) will receive a homologous transfusion.

DETAILED DESCRIPTION:
Homologous blood transfusions (HBT) and autologous blood transfusions (ABT) are abused by athletes to illegally increase their hemoglobin mass and subsequently improve oxygen transport.

Anti-Doping labs use flow-cytometry to detect HBT in cheating athletes, but athletes avoid being tested positive by matching their blood for minor blood groups before transfusion. Recent publications suggest that DNA typing by Capillary Electrophoresis or RT-PCR might be an alternative way to detect this kind of doping in athletes. Unfortunately, no data exist on the clearance of DNA after transfusion of one bag of blood using this methodology.

For the detection of doping with ABT, there is no direct method available and only the biological passport, a longitudinal collection of hematological parameters can indicate doping. Recently RBC Microparticles (RBC-MPs) have been described as a potential biomarker for autologous transfusion. However, also for this methodology, no data on the clearance time of RBC-MPs are available.

Thus, in this World Anti-Doping Agency (WADA) approved and sponsored project. The investigators plan to perform a clinical trial in which six healthy subjects receive an ABT and six healthy subjects or patients a HBT. Blood samples will be collected before and at several time-points after transfusion. For the detection of HBT the samples will be analyzed by the official method (cytometry), and the two genotyping methods (STR and RT-PCR) to compare these different techniques and to see if DNA-typing can replace cytometry.

For the ABT the collected samples will be analyzed for RBC-MPs on a cytometer dedicated for Microparticles.

ELIGIBILITY:
Inclusion Criteria:

* both genders,
* age 20-50 years and
* preferably physically active but no elite athletes subjected to Anti-Doping testing.

Exclusion Criteria:

* vulnerable subjects
* not willing to participate
* not signing the ICF
* patients with end-organ failure

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Donor DNA (# of loci with triplets or quadruplets): | 12 months
  Clearance Kinetics of donor DNA which is transferred during the transfusion of one bag of homologous blood will be established.
Cellular Microparticles (10^3/uL): | 12 months
  Clearance Kinetics of cellular microparticles which are introduced during an autologous blood transfusion and are originating from red blood cells during blood storage will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Voss, Study Chair — ADLQ; Mohamed Yassin, Principal Investigator — Hamad Medical Corporation; Francesco Donati, Principal Investigator — Laboratorio Antidoping FMSI, Rome, Italy; Costas Georgakopoulos, Principal Investigator — ADLQ; Mohammed Alsayrafi, Principal Investigator — ADLQ; Jean-Charles Grivel, Principal Investigator — Sidra Medicine; Christophe Raynaud, Principal Investigator — Sidra Medicine
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Background] Voss SC, Thevis M, Schinkothe T, Schanzer W. Detection of homologous blood transfusion. Int J Sports Med. 2007 Aug;28(8):633-7. doi: 10.1055/s-2007-965076. Epub 2007 Jul 5. PMID 17614019
- [Background] Giraud S, Robinson N, Mangin P, Saugy M. Scientific and forensic standards for homologous blood transfusion anti-doping analyses. Forensic Sci Int. 2008 Jul 18;179(1):23-33. doi: 10.1016/j.forsciint.2008.04.007. Epub 2008 Jun 2. PMID 18514452
- [Background] Krotov G, Nikitina M, Rodchenkov G. Possible cause of lack of positive samples on homologous blood transfusion. Drug Test Anal. 2014 Nov-Dec;6(11-12):1160-2. doi: 10.1002/dta.1736. Epub 2014 Oct 20. PMID 25331764
- [Background] Donati F, Stampella A, de la Torre X, Botre F. Investigation on the application of DNA forensic human identification techniques to detect homologous blood transfusions in doping control. Talanta. 2013 Jun 15;110:28-31. doi: 10.1016/j.talanta.2013.02.042. Epub 2013 Mar 18. PMID 23618171
- [Background] Stampella A, Di Marco S, Pirri D, de la Torre X, Botre F, Donati F. Application of DNA-based forensic analysis for the detection of homologous transfusion of whole blood and of red blood cell concentrates in doping control. Forensic Sci Int. 2016 Aug;265:204-10. doi: 10.1016/j.forsciint.2016.04.021. Epub 2016 Apr 30. PMID 27175858
- [Background] Manokhina I, Rupert JL. A DNA-based method for detecting homologous blood doping. Anal Bioanal Chem. 2013 Dec;405(30):9693-701. doi: 10.1007/s00216-013-7122-8. Epub 2013 Jul 11. PMID 23842898
- [Background] Alizadeh M, Bernard M, Danic B, Dauriac C, Birebent B, Lapart C, Lamy T, Le Prise PY, Beauplet A, Bories D, Semana G, Quelvennec E. Quantitative assessment of hematopoietic chimerism after bone marrow transplantation by real-time quantitative polymerase chain reaction. Blood. 2002 Jun 15;99(12):4618-25. doi: 10.1182/blood.v99.12.4618. PMID 12036896
- [Background] Ni W, Le Guiner C, Moullier P, Snyder RO. Development and utility of an internal threshold control (ITC) real-time PCR assay for exogenous DNA detection. PLoS One. 2012;7(5):e36461. doi: 10.1371/journal.pone.0036461. Epub 2012 May 3. PMID 22570718
- [Background] Almizraq RJ, Seghatchian J, Acker JP. Extracellular vesicles in transfusion-related immunomodulation and the role of blood component manufacturing. Transfus Apher Sci. 2016 Dec;55(3):281-291. doi: 10.1016/j.transci.2016.10.018. Epub 2016 Oct 28. PMID 27865649
- [Background] Straat M, Boing AN, Tuip-De Boer A, Nieuwland R, Juffermans NP. Extracellular Vesicles from Red Blood Cell Products Induce a Strong Pro-Inflammatory Host Response, Dependent on Both Numbers and Storage Duration. Transfus Med Hemother. 2016 Jul;43(4):302-305. doi: 10.1159/000442681. Epub 2015 Dec 16. PMID 27721707
- [Background] van der Pol E, Coumans FA, Grootemaat AE, Gardiner C, Sargent IL, Harrison P, Sturk A, van Leeuwen TG, Nieuwland R. Particle size distribution of exosomes and microvesicles determined by transmission electron microscopy, flow cytometry, nanoparticle tracking analysis, and resistive pulse sensing. J Thromb Haemost. 2014 Jul;12(7):1182-92. doi: 10.1111/jth.12602. Epub 2014 Jun 19. PMID 24818656
- [Background] Nielsen MH, Beck-Nielsen H, Andersen MN, Handberg A. A flow cytometric method for characterization of circulating cell-derived microparticles in plasma. J Extracell Vesicles. 2014 Feb 4;3. doi: 10.3402/jev.v3.20795. eCollection 2014. PMID 24511371
- [Background] Rubin O, Crettaz D, Tissot JD, Lion N. Pre-analytical and methodological challenges in red blood cell microparticle proteomics. Talanta. 2010 Jun 30;82(1):1-8. doi: 10.1016/j.talanta.2010.04.025. Epub 2010 Apr 22. PMID 20685428
- [Background] Rank A, Nieuwland R, Crispin A, Grutzner S, Iberer M, Toth B, Pihusch R. Clearance of platelet microparticles in vivo. Platelets. 2011;22(2):111-6. doi: 10.3109/09537104.2010.520373. Epub 2011 Jan 13. PMID 21231854
- [Background] Voss SC, Jaganjac M, Al-Thani AM, Grivel JC, Raynaud CM, Al-Jaber H, Al-Menhali AS, Merenkov ZA, Alsayrafi M, Latiff A, Georgakopoulos C. Analysis of RBC-microparticles in stored whole blood bags - a promising marker to detect blood doping in sports? Drug Test Anal. 2017 Nov;9(11-12):1794-1798. doi: 10.1002/dta.2212. Epub 2017 Jun 20. PMID 28474406